CLINICAL TRIAL: NCT06670677
Title: OBPM_FORESEE2024: Evaluation of the Clinical Benefit of the Aktiia Blood Pressure Monitoring for Early Awareness of Hypertension and Prediction of Cardiovascular Risk in a Multi-ethnic European Population: an Observational Cohorts' Study
Brief Title: Evaluation of the Clinical Benefit of the Aktiia Blood Pressure Monitoring for Early Awareness of Hypertension and Prediction of Cardiovascular Risk
Acronym: FORESEE2024
Status: Recruiting | Type: Observational
Sponsor: Aktiia SA (Industry)
Responsible Party: Sponsor
Other Study IDs: OBPM_FORESEE2024; SNCTP (Other: KOFAM)
Record Dates: First submitted 2024-10-23; First posted 2024-11-01 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Cardiovascular Risk; Blood Pressure Check (Hypertension Screening)
Keywords: hypertension; blood pressure; Hypertensive; cardiovascular diseases; cardiovascular risk; prediction
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ARM 1 G1 Aktiia users Android: Research participants are Aktiia G1 users with Android operating system, i.e. individuals who already purchased the Aktiia G1 device out of the context of the study, located in Switzerland, Germany or UK, and owning a smartphone with Android operating system.
  Interventions: Other: Lifestyle survey completion; Other: Unlimited on-demand blood pressure measurements with G2C; Other: Continual blood pressure measurements with G1
- ARM 2 G1 AKTIIA users iOS: Research participants are Aktiia G1 users with iOS operating system, i.e. individuals who already purchased the Aktiia G1 device out of the context of the study, located in Switzerland, Germany or UK, and owning a smartphone with iOS operating system.
  Interventions: Other: Lifestyle survey completion; Other: Unlimited on-demand blood pressure measurements with G2C; Other: Continual blood pressure measurements with G1
- ARM 3 non-Aktiia-G1-users Android & iOS: Research participants are non-Aktiia-G1 users (they do not own an Aktiia G1 device at their inclusion in the study), located in Switzerland, Germany or UK, and owning a smartphone with either iOS or Android operating system.
  Interventions: Other: Lifestyle survey completion; Other: Unlimited on-demand blood pressure measurements with G2C

INTERVENTIONS:
Other: Lifestyle survey completion — For the next 10 years, starting at their inclusion in the research project and every 6 months thereafter: fill in an online survey on their lifestyle- health- socioeconomic environment. The completion of a survey lasts 5min maximum.
Other: Unlimited on-demand blood pressure measurements with G2C — For the next 10 years: take unlimited on-demand measurements with the Aktiia G2C feature (finger measurement) while seated
Other: Continual blood pressure measurements with G1 — For the next 10 years: wear their 24/7 Aktiia G1 device continuously as they would outside the context of the research project.
  Groups: ARM 1 G1 Aktiia users Android; ARM 2 G1 AKTIIA users iOS

SUMMARY:
Because Aktiia S.A. has been the first-ever company to put in the market an Optical Blood Pressure Monitoring device, there is a need for Aktiia S.A. to correlate for the first time continual Blood Pressure monitoring and the evolution of environmental and health factors to improve hypertension management.

DETAILED DESCRIPTION:
ARM 1:

N1~ 3'300 subjects.

Research participants are Aktiia G1 users with Android operating system, i.e. individuals who already purchased the Aktiia G1 device out of the context of the study, located in Switzerland, Germany or UK, and owning a smartphone with Android operating system. ARM 1 research participants are asked to:

* For the next 10 years: wear their 24/7 Aktiia G1 device continuously as they would outside the context of the research project,
* For the next 10 years, starting at their inclusion in the research project and every 6 months thereafter: fill in an online survey on their lifestyle- health- socioeconomic environment.
* Additionally, once the Aktiia One App is released and for the next 10 years:
* Take an on-demand measurement with the Aktiia G2C feature (finger measurement) while seated.

ARM 2:

N2~ 6'600 subjects.

Research participants are Aktiia G1 users with iOS operating system, i.e. individuals who already purchased the Aktiia G1 device out of the context of the study, located in Switzerland, Germany or UK, and owning a smartphone with iOS operating system. ARM 2 research participants are asked to:

* For the next 10 years: wear their 24/7 Aktiia G1 device continuously as they would outside the context of the research project,
* For the next 10 years, starting at their inclusion in the research project and every 6 months thereafter: fill in an online survey on their lifestyle- health- socioeconomic environment. The completion of a survey lasts 5min maximum.
* Additionally, once the Aktiia One App is released and for the next 10 years:
* Take an on-demand measurement with the Aktiia G2C feature (finger measurement) while seated.

ARM 3:

N3~ 5'000 subjects.

Research participants are non-Aktiia-G1 users (they do not own an Aktiia G1 device at their inclusion in the study), located in Switzerland, Germany or UK, and owning a smartphone with either iOS or Android operating system. ARM 3 research participants are asked to:

* For the next 10 years, starting at their inclusion in the research project and every 6 months thereafter: fill in an online survey on their lifestyle- health- socioeconomic environment. The completion of a survey lasts 5min maximum.
* At their inclusion in the study: download the Aktiia One App to access G2C functionality with on-demand measurements at fingertip using the smartphone's camera.
* For the next 10 years, starting at their inclusion in the research project and thereafter:

  * Take unlimited on-demand measurements with the Aktiia G2C feature.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 21 to 85 years old
2. Subjects living in Switzerland, Germany or in the UK
3. Subjects that are:

   Aktiia users owning a smartphone with either iOS or Android operating system (ARMs 1 and 2); or Aktiia non-users owning a smartphone with iOS or Android operating system (ARM 3)
4. Subjects agreeing to follow the study procedures.

Exclusion Criteria:

1. Subjects suffering from sustained cardiac arrhythmias that can lead to weak or unstable pressure pulses including resting tachycardia (heart rate at rest > 120bpm) and atrial fibrillation;
2. Subjects suffering from pathologies that systematically reduce peripheral perfusion including Raynaud's disease, diabetes, renal dysfunctions (eGFR < 30mL / min / 1.73 m2), untreated hyper-/ hypothyroidism, pheochromocytoma, or arteriovenous fistula;
3. Subjects suffering from polyneuropathy;
4. on pregnant women;
5. Subjects with damaged / injured skin at the wrists (for bracelet measurements) or at index fingers (for camera measurements)
6. Subjects with amputated index fingers (for camera measurements) or amputated upper limb;
7. Subjects below 21 years old and above 85 years old.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any subjects that respect the study inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2035-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
Multivariate models relating data from 24/7 Aktiia the G1 device continual BP monitoring with sociodemographic - lifestyle - and health factors | 10 years
  Strength and direction of the correlation coefficient between continuous blood pressure readings and various survey-derived factors such as sociodemographic variables, lifestyle habits, and health metrics.

SECONDARY OUTCOMES:
Global scale projections of the benefit of the early awareness of hypertension with the spot-check Aktiia G2C device at the fingertip | 10 years
  Proportion of subjects with early hypertension awareness enabled by the fingertip spot-check feature of the Aktiia G2C device.

CONTACTS AND LOCATIONS:
Locations (2):
- Fully remote study- no physical investigational site, Lausanne, Switzerland
- Fully remote study- no physical investigational site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No